CLINICAL TRIAL: NCT01869894
Title: A Prospective Randomized Study for Efficacy of Uncovered Double Bare Metallic Stent Compared to Uncovered Single Bare Metallic Stent in Malignant Biliary Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2013-0204
Record Dates: First submitted 2013-05-29; First posted 2013-06-05 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Malignant Biliary Obstruction
Keywords: Malignant biliary obstruction; metal stent; patency

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- uncovered double bare metallic stent (S&G Biotech.) (Active Comparator): uncovered double bare metallic stent
  Interventions: Procedure: metallic biliary stent insertion (double bare - S&G Biotech.)
- uncovered single bare metallic stent (S&G Biotech.) (Active Comparator): uncovered single bare metallic stent
  Interventions: Procedure: metallic biliary stent insertion (single bare - S&G Biotech.)
- uncovered single bare metallic stent (Taewoong Medical.) (Active Comparator): uncovered single bare metallic stent
  Interventions: Procedure: metallic biliary stent insertion (single bare - Taewoong Medical.)

INTERVENTIONS:
Procedure: metallic biliary stent insertion (double bare - S&G Biotech.) — The patients who had malignant biliary obstruction will be enrolled our study. Enrolled patient will be randomized to three group (uncovered double bare metallic stent (S&G Biotech.) vs. uncovered single bare metallic stent (S&G Biotech.) vs. uncovered single bare metallic stent (Taewoong Medical.)). After metallic biliary stent insertion, enrolled patients will be followed at least one time per one month. Blood test (including total bilirubin, gamma-GT) will be done for follow-up study. During follow-up period, if biliary obstruction is suspected, imaging study (CT or MRCP) will be done. With such follow-up tools, we compare 6-month patency rate and median patency duration among three groups.
  Arms: uncovered double bare metallic stent (S&G Biotech.)
Procedure: metallic biliary stent insertion (single bare - S&G Biotech.) — The patients who had malignant biliary obstruction will be enrolled our study. Enrolled patient will be randomized to three group (uncovered double bare metallic stent (S&G Biotech.) vs. uncovered single bare metallic stent (S&G Biotech.) vs. uncovered single bare metallic stent (Taewoong Medical.)). After metallic biliary stent insertion, enrolled patients will be followed at least one time per one month. Blood test (including total bilirubin, gamma-GT) will be done for follow-up study. During follow-up period, if biliary obstruction is suspected, imaging study (CT or MRCP) will be done. With such follow-up tools, we compare 6-month patency rate and median patency duration among three groups.
  Arms: uncovered single bare metallic stent (S&G Biotech.)
Procedure: metallic biliary stent insertion (single bare - Taewoong Medical.) — The patients who had malignant biliary obstruction will be enrolled our study. Enrolled patient will be randomized to three group (uncovered double bare metallic stent (S&G Biotech.) vs. uncovered single bare metallic stent (S&G Biotech.) vs. uncovered single bare metallic stent (Taewoong Medical.)). After metallic biliary stent insertion, enrolled patients will be followed at least one time per one month. Blood test (including total bilirubin, gamma-GT) will be done for follow-up study. During follow-up period, if biliary obstruction is suspected, imaging study (CT or MRCP) will be done. With such follow-up tools, we compare 6-month patency rate and median patency duration among three groups.
  Arms: uncovered single bare metallic stent (Taewoong Medical.)

SUMMARY:
Our study is the prospective randomized study for efficacy of uncovered double bare metallic stent compared to uncovered single bare metallic stent in malignant biliary obstruction

ELIGIBILITY:
Inclusion Criteria:

* The patients who had malignant biliary obstruction

Exclusion Criteria:

* The patients who had resectable biliary malignancy
* The patients who had hilar obstruction
* The patients who had duodenal obstruction
* The patients who had other malignancy which is not related to biliary obstruction
* The patients who had uncontrolled infection
* The patients who had poor performance (ECOG =3 or 4)
* The patients who were not acquired informed consent
* The patients who had technically difficult structure for ERCP

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Median patency duration | Approximately 6 months later since the date of stent insertion
  Primary end point : A. Median patency duration

SECONDARY OUTCOMES:
6-months patency rate | Approximately 6 months later since the date of stent insertion
  Secondary end point : A. 6-months patency rate

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

REFERENCES:
- [Result] Isayama H, Komatsu Y, Tsujino T, Sasahira N, Hirano K, Toda N, Nakai Y, Yamamoto N, Tada M, Yoshida H, Shiratori Y, Kawabe T, Omata M. A prospective randomised study of "covered" versus "uncovered" diamond stents for the management of distal malignant biliary obstruction. Gut. 2004 May;53(5):729-34. doi: 10.1136/gut.2003.018945. PMID 15082593
- [Result] Davids PH, Groen AK, Rauws EA, Tytgat GN, Huibregtse K. Randomised trial of self-expanding metal stents versus polyethylene stents for distal malignant biliary obstruction. Lancet. 1992 Dec 19-26;340(8834-8835):1488-92. doi: 10.1016/0140-6736(92)92752-2. PMID 1281903
- [Derived] Lee HJ, Chung MJ, Park JY, Park SW, Nam CM, Song SY, Bang S. A prospective randomized study for efficacy of an uncovered double bare metal stent compared to a single bare metal stent in malignant biliary obstruction. Surg Endosc. 2017 Aug;31(8):3159-3167. doi: 10.1007/s00464-016-5341-8. Epub 2016 Nov 18. PMID 27864713